CLINICAL TRIAL: NCT04885647
Title: A Multicenter, Randomized, Open-label, Phase 2 Study of YPEG-rhEPO in Patients Suffered From Anemia Due to Chronic Kidney Disease, Who Has Previously Treated With rhEPO and Maintains the Hemoglobin in a Stabilize State
Brief Title: A Study of YPEG-rhEPO in Patients Suffered From Anemia Due to Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TB1901EPO
Record Dates: First submitted 2021-05-08; First posted 2021-05-13 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Renal Anemia of Chronic Kidney Disease
Keywords: YPEG rhEPO; rhEPO; erythropoietin; anemia; dialysis; hemodialysis; chronic kidney disease
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm1 (Experimental): Low dose once every 2 weeks group
  Interventions: Drug: YPEG-rhEPO
- Arm2 (Experimental): Low dose once every 4 weeks group
  Interventions: Drug: YPEG-rhEPO
- Arm3 (Experimental): High dose once every 2 weeks group
  Interventions: Drug: YPEG-rhEPO
- Arm4 (Experimental): High dose once every 4 weeks group
  Interventions: Drug: YPEG-rhEPO

INTERVENTIONS:
Drug: YPEG-rhEPO — YPEG-rhEPO，low dose，were subcutaneous injected once every two weeks for 13 weeks.
  Arms: Arm1
Drug: YPEG-rhEPO — YPEG-rhEPO，low dose，were subcutaneous injected once every four weeks for 13 weeks.
  Arms: Arm2
Drug: YPEG-rhEPO — YPEG-rhEPO, high dose，were subcutaneous injected once every two weeks for 13 weeks.
  Arms: Arm3
Drug: YPEG-rhEPO — YPEG-rhEPO，high dose，were subcutaneous injected once every four weeks for 13 weeks.
  Arms: Arm4

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of YPEG rhEPO, a recombinant human erythropoietin pegylated by Y shape polyethylene glycol, in patients with anemia due to Chronic Kidney Disease (CKD), assessed by hemoglobin maintenance, adverse events and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years old, including 18 and 70 years.
* Subjects who are diagnosed of chronic kidney disease and receiving hemodialysis (KT/V greater than or equal to 1.2). And those who had received hemodialysis, performed 2 to 3 times a week and 4 to 5 hours for every dialysis, for at least 12 weeks prior to deliver of YPEG-EPO.
* Subjects receiving rhEPO treatment, including subcutaneous and intravenous injection, for anemia due to chronic kidney disease for at least 12 weeks before randomized. And in addition, the serum hemoglobin should keep stable during the previous 12 weeks, which was defined as serum hemoglobin obtained from tests taken once a month (once a month means at least 4 weeks interval between two tests) were always kept between 100g/L and 120g/L, or else mean hemoglobin of two different tests, which were taken at least 4 weeks apart, is between 100g/L and 120g/L.
* Transferrin saturation (TSAT) greater than 20% or serum ferritin (SF) greater than 200ng/mL, serum folate greater or equal to the lower normal limit (ULN), serum vitamin B12 greater or equal to ULN，before enrollment.
* Understand and sign the informed consent form voluntarily.

Exclusion Criteria:

* Women of pregnancy, lactating, or planning to pregnant, or patients who are planning to donate sperms/eggs during the study period.
* Subjects who are allergic to rhEPO or any of its components, or with any other evidenced allergy history that make it not suitable for participation.
* Subjects who are receiving Roxadustat Capsules at screening.
* Anemia caused by diseases or causes other than CKD, such as bleeding, hemolysis, vitamin or folate deficiency. Obvious bleeding evidence that requires blood transfusion during the lead-in period.
* Subjects suffering from pure red-cell anemia (PRCA) according to previously erythropoietin treatment.
* Subjects with serious disease or function deficiency in major organ/system, such as：

  1. Medical history of myocardial infarction, cerebral stroke, vascular access thrombosis, or pulmonary embolism. Combined congestive heart failure (NYHA cardiac function equal to or grade than III). Hypertensions poorly controlled by medication (systolic blood pressure higher than 170mmHg and/or diastolic blood pressure higher than 100mmHg), or postural hypotension (systolic blood pressure below 90mmHg).
  2. Medical history of malignancy, hematological disease, obvious bleeding disease, epilepsy, neuropsychiatric disease, or family history of neuropsychiatric disease.
  3. Poorly controlled autoimmune diseases (including but not limit to systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, autoimmune thrombocytopenia).
  4. Poorly controlled endocrine diseases, (including but not limit to thyroid disease, parathyroid disease, diabetes mellitus).
  5. Co-infected with HAV, HBV, HCV, HIV, Syphilis, etc..
  6. Currently suffering from severe infection or inflammation (C-reactive protein greater than 30mg / L), or currently receiving antibiotics.
* Red blood cell count greater than 6.0×10^12/L for men while greater than 5.5×10^12/L for female; Platelets greater than 500×10^9/L; serum albumin lower than 30g/L; Alanine aminotransferase higher than 2 ULN, aspartame aminotransferase higher than 2ULN; Parathyroid hormone greater than 800pg/mL.
* Subjects who plan to undergo coronary artery bypass grafting (CABG), to undergo orthopedic surgery, to receive kidney transplantation, or to undergo any other major operation during the study period.
* Drug addicts or alcoholics.
* Vascular malformations (such as internal jugular vein malformation) makes it inappropriately for Hemodialysis catheterization.
* Expected survival of a certain subject is less than 12 months.
* Subjects participated in any other clinical trial within 3 months prior to screening.
* Any other situation that is not suitable for participation in this study according to the investigator's judgment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Changes of mean hemoglobin compared to baseline. | 14 weeks for every two weeks groups, and 16 weeks for every four weeks groups.

SECONDARY OUTCOMES:
Proportion of patients with hemoglobin keeping within the target range (the target hemoglobin range is defined as hemoglobin keeping between 100g/L and 120g/L). | 14 weeks for every two weeks groups, and 16 weeks for every four weeks groups.
Proportion of patients with hemoglobin fluctuations within ±10g/L compared to baseline. | 14 weeks for every two weeks groups, and 16 weeks for every four weeks groups.
Mean time of hemoglobin keeping within the target range. | 14 weeks for every two weeks groups, and 16 weeks for every four weeks groups.
Mean time from baseline to the first dose adjustment. | 14 weeks for every two weeks groups, and 16 weeks for every four weeks groups.
Changes of hemoglobin compared to baseline at the time of first dose adjustment. | 14 weeks for every two weeks groups, and 16 weeks for every four weeks groups.
Proportion of patients with dose adjustment. | 14 weeks for every two weeks groups, and 16 weeks for every four weeks groups.
Proportion of patients requiring blood transfusion. | 14 weeks for every two weeks groups, and 16 weeks for every four weeks groups.

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Beijing Anzhen Hospital,Capital Medical University, Beijing, Beijing Municipality
  - The Second Affiliated Hospital Of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital Of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat sen University, Guanzhou, Guangdong
  - Renmin Hospital of Wuhan University/Hubei General Hospital, Wuhan, Hubei
  - The Third Xiangya Hospital Of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First Affiliated Hospital Of Baotou Medical college,Inner Mongolia University Of Science and Technology, Hohhot, Inner Mongol
  - Huai'an Second People's Hospital/The Affiliated Huaian Hospital Of Xuzhou Medical University, Huai'an, Jiangsu
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - Xi'an Gaoxin Hospital, Xi’an, Shanxi
  - The First Affiliated Hospital Of Chengdu Medical college, Chengdu, Sichuan
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Lishui Municipal Central Hospital, Lishui, Zhejiang

IPD SHARING:
Plan to Share IPD: No